CLINICAL TRIAL: NCT01998828
Title: A Phase 2, Open-label, Randomized Study to Evaluate the Safety and Efficacy of Momelotinib in Subjects With Polycythemia Vera or Essential Thrombocythemia
Brief Title: Safety and Efficacy of Momelotinib in Subjects With Polycythemia Vera or Essential Thrombocythemia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Sierra Oncology LLC - a GSK company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-354-0101; 2013-004105-11 (EudraCT Number)
Record Dates: First submitted 2013-11-25; First posted 2013-12-02 (Estimated); Last update posted 2020-04-20 (Actual); Status verified 2020-04

CONDITIONS: Polycythemia Vera; Essential Thrombocythemia
Keywords: Polycythemia; Polycythemia Vera; Essential Thrombocythemia; Thrombocytosis; Myeloproliferative Disorders; Bone Marrow Diseases; Hematologic Diseases; Blood Coagulation Disorders; Blood Platelet Disorders; Hemorrhagic Disorders
MeSH Terms: conditions — Polycythemia Vera; Thrombocythemia, Essential; Polycythemia; Thrombocytosis; Myeloproliferative Disorders; Bone Marrow Diseases; Hematologic Diseases; Blood Coagulation Disorders; Blood Platelet Disorders; Hemorrhagic Disorders | interventions — N-(cyanomethyl)-4-(2-((4-(4-morpholinyl)phenyl)amino)-4-pyrimidinyl)benzamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Momelotinib 100 mg PV (Experimental): Participants with polycythemia vera will receive 100 mg of momelotinib.
  Interventions: Drug: Momelotinib
- Momelotinib 200 mg PV (Experimental): Participants with polycythemia vera will receive 200 mg of momelotinib.
  Interventions: Drug: Momelotinib
- Momelotinib 100 mg ET (Experimental): Participants with essential thrombocythemia will receive 100 mg of momelotinib.
  Interventions: Drug: Momelotinib
- Momelotinib 200 mg ET (Experimental): Participants with essential thrombocythemia will receive 200 mg of momelotinib.
  Interventions: Drug: Momelotinib

INTERVENTIONS:
Drug: Momelotinib — Momelotinib tablet administered orally once daily
  Other Names: GS-0387; CYT387

SUMMARY:
This open-label study is to determine the safety and efficacy of momelotinib in participants with either polycythemia vera (PV) or essential thrombocythemia (ET) who have not yet received treatment with a Janus kinase (JAK) inhibitor.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of either PV or ET as defined by the 2008 World Health Organization (WHO) Diagnostic Criteria
* Requires treatment for PV or ET, in the opinion of the study investigator
* Intolerant of, resistant to, or refuses current or available treatment for PV or ET
* Direct bilirubin ≤ 2.0 x upper limit of the normal range (ULN)
* Aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 3 x ULN
* Calculated creatinine clearance (CrCl) of ≥ 45 mL/min
* Life expectancy > 24 weeks
* Male subjects and female subjects of childbearing potential who engage in heterosexual intercourse must agree to use protocol specified method(s) of contraception
* Females who are nursing must agree to discontinue nursing before the first dose of study drug
* Able to comprehend and willing to sign informed consent form

Exclusion Criteria:

* Prior splenectomy
* Uncontrolled intercurrent illness, per protocol
* Known positive status for human immunodeficiency virus (HIV)
* Chronic active or acute viral hepatitis A, B, or C infection, or hepatitis B or C carrier
* Myeloproliferative neoplasm-directed therapy, other than aspirin, hydroxyurea, anagrelide, and/or phlebotomy, within 21 days prior to the first dose of study drug
* Anagrelide within 7 days prior to the first dose of study drug
* Presence of peripheral neuropathy ≥ Grade 2
* Unwilling or unable to take oral medication
* Prior use of a JAK1 or JAK2 inhibitor
* Use of strong CYP3A4 inducers within 1 week prior to the first dose of study drug
* QTc interval > 450 msec, unless attributed to bundle branch block

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2014-02-19 (Actual); Primary Completion 2015-03-17 (Actual); Study Completion 2015-05-07 (Actual)

PRIMARY OUTCOMES:
Overall response rate | Up to 24 weeks
  For the PV Cohort, overall response rate (ORR) is defined as the proportion of participants with all of the following at some point during the treatment period:
  * Hematocrit < 45% in the absence of phlebotomy that lasts at least 4 weeks
  * White blood cell (WBC) count < 10 x 10^9/L that lasts at least 4 weeks
  * Platelet count ≤ 400 x 10^9/L that lasts at least 4 weeks
  * Resolution of palpable splenomegaly that lasts at least 4 weeks
  For the ET Cohort, overall response rate is defined as the proportion of participants with all of the following at some point during the treatment period:
  * WBC count < 10 x 10^9/L that lasts at least 4 weeks
  * Platelet count ≤ 400 x 10^9/L that lasts at least 4 weeks
  * Resolution of palpable splenomegaly that lasts at least 4 weeks

SECONDARY OUTCOMES:
Confirmed overall response rate | Up to 24 weeks
  Confirmed overall response rate is defined as the proportion of participants who meet all the criteria listed for the primary endpoints of PV or ET, sustained for at least 12 weeks.
Proportion of participants with hematocrit < 45% in the absence of phlebotomy that lasts at least 4 weeks | Up to 24 weeks
Proportion of participants with WBC < 10 x 10^9/L that lasts at least 4 weeks | Up to 24 weeks
Proportion of participants with platelet count ≤ 400 x 10^9/L that lasts at least 4 weeks | Up to 24 weeks
Proportion of participants with resolution of palpable splenomegaly that lasts at least 4 weeks | Up to 24 weeks
Proportion of participants with ≥ 10 point decrease in modified Myeloproliferative Neoplasm Symptom Assessment Form Total Symptom Score (MPNSAF TSS) compared to baseline that lasts at least 12 weeks | Up to 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Peter Lee, MD, PhD, Study Director — Gilead Sciences
Locations (15):
- United States (5):
  - Scottsdale, Arizona
  - Whittier, California
  - Tupelo, Mississippi
  - St Louis, Missouri
  - Houston, Texas
- Australia (2):
  - Frankston, Victoria
  - Parkville, Victoria
- Canada (3):
  - Vancouver, British Columbia
  - Toronto, Ontario
  - Montreal, Quebec
- France (3):
  - La Tronche
  - Nantes
  - Paris
- Germany (2):
  - Dresden
  - Minden

REFERENCES:
- [Derived] Verstovsek S, Courby S, Griesshammer M, Mesa RA, Brachmann CB, Kawashima J, Maltzman JD, Shao L, Xin Y, Huang D, Bajel A. A phase 2 study of momelotinib, a potent JAK1 and JAK2 inhibitor, in patients with polycythemia vera or essential thrombocythemia. Leuk Res. 2017 Sep;60:11-17. doi: 10.1016/j.leukres.2017.05.002. Epub 2017 May 30. PMID 28622623